CLINICAL TRIAL: NCT06372665
Title: Safety Observation of the Vero Cell-derived Inactivated Japanese Encephalitis Vaccine (JEV-I) Given With Primary Immunization in a Large Amount of Healthy Children Aged 8 Months and Older
Brief Title: Safety Observation of the Japanese Encephalitis Vaccine Given With a Primary Immunization
Status: Completed | Type: Observational
Sponsor: Liaoning Chengda Biotechnology CO., LTD (Industry)
Responsible Party: Sponsor
Other Study IDs: CDB-IV-JE-025202301
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Japanese Encephalitis
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Vero Cell-derived Inactivated Japanese Encephalitis Vaccine Group: Healthy children aged 8 months and above who choose to receive the study vaccine for primary immunization at their own expense in Jiangsu Province

SUMMARY:
This is a single-arm, non-randomized, open-label post-marketing safety observation study. The purpose of this study is to investigate the safety of JEV-I given with primary immunization in a large amount of healthy children aged 8 months and older.

DETAILED DESCRIPTION:
Healthy children aged 8 months and older who choose to receive the study vaccine for primary immunization at their own expense in Jiangsu Province will be invited to participate in this study. No study vaccine will be supplied or administered as part of this study, participants will be monitored following vaccine administration in clinical settings.

The primary immunization program with JEV-I requires 2 intramuscular doses administered 7-10 days apart. All participants will be observed for the incidence of any adverse events (AEs) within 30 minutes and from 30 minutes to 7 days after each vaccination, including local and systemic reactions. Additionally, all participants will be observed for unsolicited AEs within 30 days after after each vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children who have received the inactivated Japanese encephalitis vaccine.
* Legal guardian of the participants voluntarily participates in the clinical trial and signs an informed consent form.
* Legal guardian of the subject has the ability to understand the procedures of the study and accept all scheduled visits.

Exclusion Criteria:

-

Min Age: 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy children aged 8 months and older who voluntarily receive the research vaccines within Jiangsu Province
Sampling Method: Non-Probability Sample
Enrollment: 15357 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants Reporting Solicited Local and Systemic Adverse Events, and Unsolicited Adverse Events | 30 days following each vaccination
  Adverse events (AEs) are defined as all adverse medical events that occur in participants after receiving the investigational drug, which can manifest as symptoms, signs, diseases, or abnormal laboratory tests, but they may not necessarily have a causal relationship with the investigational drug.
  Unsolicited AEs will be collected within 30 days after each dose of vaccine administration, while solicited adverse reactions will be collected within 30 minutes and 30 minutes to 7 days after each dose of vaccine administration. A structured form (pre-listed) will be used to record the local and systemic reactions collected below.
  Local reactions:
  * Pain
  * Induration
  * Ecchymosis (Redness)
  * Pruritus
  * Rash
  Systemic reactions:
  * Headache
  * Courbature (not from injection site)
  * Diarrhea
  * Dysphagia
  * Anorexia
  * Vomiting
  * Sickness
  * Cough
  * Dyspnea
  * Irritability
  * Sleepiness
  * Acute allergic reaction
  * Pain (not from injection site)

CONTACTS AND LOCATIONS:
Overall Officials: Huanyu Wang, Study Director — Liaoning Chengda Biotechnology CO., LTD
Locations (1):
- Jiangsu Provincial Center for Disease Control and Prevention, Nanjing, Jiangsu, China